CLINICAL TRIAL: NCT05806411
Title: Calcific Aortic Valve Disease: a Multidisciplinary Approach to Investigate the Role of Bacteria as Trigger of a Chronic Inflammation in the Pathogenesis of Calcification
Brief Title: Calcific Aortic Valve Disease:the Role of Bacteria as Trigger of a Chronic Inflammation
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: University of Pavia (Other)
Responsible Party: Sponsor
Other Study IDs: CAvD
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Calcific Aortic Valve Diasease
Keywords: Calcific aortic valve disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Total calcium content will be analyzed from cusps explants upon tissue homogenization, metal chelation and spectroscopic quantification qPCR, using RNA extracted from a section of the samples described above, will be used to determine the tissue expression of early and late osteogenic markers.
  For bacteria detection an aliquot of the valve tissue will be minced and homogenized in phosphate saline solution for genomic DNA extraction. The approach that we propose is based on a pan bacterial PCR amplifying 16S rDNA, followed by the sequencing of V1-V3 regions of 16S rDNA through Illumina technology for all the samples proved to be positive for the pan bacterial PCR.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with calcific aortic sclerosis (stage III and IV) that are going to be treated with traditional surgery according to International Guidelines will be enrolled as cases.
  Interventions: Diagnostic Test: Analysis of calcific aortic valves
- Controls: Patients that will undergo a cardiac transplantation (for nonvalvular cardiac disease) or patients with aortic valve insufficiency will be enrolled as controls
  Interventions: Diagnostic Test: Analysis of calcific aortic valves

INTERVENTIONS:
Diagnostic Test: Analysis of calcific aortic valves — Microbiologic analysis of calcofic aortic valves

SUMMARY:
Calcific aoric valve disease (CAVD) is extremely common worldwide, affecting almost 50% of the population over 85 years of age, with a lethality higher than 50% at 2 years for symptomatic patients, unless aortic-valve replacement is performed. CAVD is characterized by slowly progressive fibro-calcific remodelling of the valve leaflets causing aortic stenosis. The spectrum of the disease progression starts with leaflet degeneration and progresses from early lesions to valve stenosis/obstruction, which is initially mild to moderate but eventually becomes severe. Risk factors for CAVD partly overlap those for atherosclerosis but also intake age-related tissue changes and effects of comorbiditiies (e.g. renal failure) in the overall complex mechanisms of valve leaflet degeneration, which is, at present, unpreventable, leaving aortic valve repair the only treatment option for severe aortic stenosis. In the first phase of the disease the valve becomes thickened and mildly calcified, then the disease evolves to severe valve calcification with impaired leaflet motion and vast blood flow obstruction. Calcific AS valves show advanced osteogenic metaplasia with the presence of osteoblast-like cells and chondrocytes associated with dense inflammatory infiltrates. Bacteria have been detected in the absence of diagnosis of acute infective endocarditis, but their role is still unknown. Different bacterial species (C. acnes (59%), E. faecalis (16%), S. aureus (15%), and S. pyogenes (10%)) have been typed and intramural bacterial colonization has been observed in patients with calcified structural valvular heart disease. Indeed, it has been recently demonstrated that bacterial infections can directly affect osteoblast differentiation/activation.

The Authors hypothesized that a subclinical or latent valvular bacterial infiltration facilitates a chronic inflammation and contributes to accelerated structural valve degeneration. An interdisciplinary team has been established to investigate the infective, biochemical and structural features of calcific aortic valve disease.

DETAILED DESCRIPTION:
The primary objective of the study is to dissect the bacteria contribution to valve calcification. The Authors hypothesized that a subclinical or latent valvular bacterial infiltration facilitates a chronic inflammation and contributes to accelerated structural valve degeneration. The Authors expect to find a correlation between bacterial detection (as qualitative -positive/negative, quantitative -quantitative PCR) and bone calcification markers on valves. To dissect the bacteria contribution to valve calcification, the osteogenic differentiation capabilities of primary cells obtained from cusp explanted from control and from non-calcified cusp of CAVD patients will be assessed in vitro in absence and in presence of bacterial infection. There are currently no data in the literature that can be referred to for the calculation of the sample size. Cusp calcifications do not equally affect all cusps, considering calcified cusp as cases and non-calcified cusp of the same valve as matched controls, if the probability of bacterial detection among sampled control non calcified cusps is 10% (Cohen, doi: 10.1016/S0003-4975(03)01454-1), a sample of 32 patients (with 32 calcified cusp and 96cusps) can be enrolled. This sample of 96 cusps achieves 81% power to detect an odds ratio of 5.00 versus the alternative of equal odds using a McNemar test with a 0.05 significance level. This calculation is done considering that the probability of bacterial detection in each cusp is almost independent from other cusps of the same valve (intra-valve correlation coefficient= 0.10). The Authors expect a total study duration of 24 months. The Authors estimate to complete recruitment in 12 months. The estimated primary completion is month 15 (3 months after last subject enrollment) and study completion on month 24 (12 months after last patient inclusion)

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years.
* Calcific aortic sclerosis (stage III and IV)

Exclusion Criteria:

- Inability to comply with the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with calcific aortic sclerosis (stage III and IV) that are going to be treated with traditional surgery according to International Guidelines will be enrolled as cases.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-06-18 (Estimated); Study Completion 2025-01-18 (Estimated)

PRIMARY OUTCOMES:
To analyze subclinical or latent valvular bacterial infiltration in patients with calcific aortic disease | 2 years
  Rate of bacterial infiltration in calcified and non calcified cusps and in patients and controls (co-primary endpoint) will be analysed.
To evaluate the correlation between bacterial detection (as qualitative-positive/negative-, quantitative -quantitative PCR-) and bone calcification markers on valves | 2 years
  Rate of expression of osteogenic markers and total calcium valve content in calcified and non-calcified cusps on valves of patients and controls and correlation with bacterial detection

CONTACTS AND LOCATIONS:
Overall Officials: Elena Seminari, MD, Principal Investigator — Fondazione IRCCS Policlinico San MAtteo
Locations (1):
- Fondazione IRCCS Policlinico San MAtteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Oberbach A, Schlichting N, Friedrich M, Lehmann S, Kullnick Y, Pichlmaier M, Hagl C, Bagaev E; CardiOmics group; Clinical Microbiology group; Clinical Management group. Quantification of Multiple Bacteria in Calcified Structural Valvular Heart Disease. Semin Thorac Cardiovasc Surg. 2020 Summer;32(2):255-263. doi: 10.1053/j.semtcvs.2019.10.003. Epub 2019 Oct 9. PMID 31605771
- [Background] Kwon Y, Park C, Lee J, Park DH, Jeong S, Yun CH, Park OJ, Han SH. Regulation of Bone Cell Differentiation and Activation by Microbe-Associated Molecular Patterns. Int J Mol Sci. 2021 May 28;22(11):5805. doi: 10.3390/ijms22115805. PMID 34071605
- [Background] Cohen DJ, Malave D, Ghidoni JJ, Iakovidis P, Everett MM, You S, Liu Y, Boyan BD. Role of oral bacterial flora in calcific aortic stenosis: an animal model. Ann Thorac Surg. 2004 Feb;77(2):537-43. doi: 10.1016/S0003-4975(03)01454-1. PMID 14759434
- [Result] Freeman RV, Otto CM. Spectrum of calcific aortic valve disease: pathogenesis, disease progression, and treatment strategies. Circulation. 2005 Jun 21;111(24):3316-26. doi: 10.1161/CIRCULATIONAHA.104.486738. No abstract available. PMID 15967862